CLINICAL TRIAL: NCT05625178
Title: Investigating Effects of Auricular Vagus Nerve Stimulation on Central Pain Mechanisms, Autonomic Function, and Pain Severity in People With Knee Osteoarthritis
Brief Title: Effects of Vagus Nerve Stimulation on Central Pain Sensitivity & Parasympathetic Function in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas, El Paso (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1966880-1
Record Dates: First submitted 2022-10-18; First posted 2022-11-22 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Knee Osteoarthritis; Central Pain Syndrome
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- tVNS group (Experimental): This will be a single-arm study where all study participants will receive transcutaneous vagus nerve stimulation (tVNS) at the cymba concha of the left ear for 60 minutes. The tVNS parameters will be a below-discomfort-threshold intensity with 25 Hz and a pulse width of 250 uS.
  Interventions: Device: Transcutaneous vagus nerve stimulation

INTERVENTIONS:
Device: Transcutaneous vagus nerve stimulation — tVNS will be performed by the application of an auricular electrode placed at the cymba concha of the left ear. The auricular electrode containing the anode will be applied with a conductive gel without prior disinfection. Once the electrode fits the cymba concha comfortably, the participant will lie down or take a position that is comfortable for them. Once in position, investigators initiate tVNS for 60 minutes with a below-discomfort-threshold intensity with 25 Hz and pulse width 250 uS. The electrical parameters will be modified accordingly to keep the below-discomfort threshold during the intervention.

SUMMARY:
The goal of this clinical trial is to test the feasibility and effectiveness of transcutaneous vagus nerve stimulation (tVNS) to the ear on pain and autonomic function in people with knee osteoarthritis (OA). The main questions it aims to answer are: 1) whether tVNS is feasible to be used in people with knee OA; 2) whether tVNS demonstrates the trend in improving knee pain; and 3) whether tVNS has physiological effects on autonomic function (e.g., parasympathetic function) and pain perception in the central nervous system such as brain (i.e., central pain mechanisms). Participants will be asked to complete a battery of self-reported questionnaires about their demographic and behavioral information, ethnicity, pain, sleep, psychological/emotional symptoms. Subsequently, participants will complete baseline assessment where investigators will assess their knee pain severity, central pain sensitivity, and heart rate variability (a measurement for autonomic function). Then participants will receive a 60-minute tVNS. Investigators will redo the same assessment as baseline assessment after tVNS intervention to see the degree of knee pain, central pain sensitivity, and autonomic function changes. At the end of the study, investigators will assess their satisfaction level with the tVNS intervention and the feasibility of the intervention (e.g., completion rate, side effects).

ELIGIBILITY:
Inclusion Criteria:

* chronic knee pain consistent with a clinical osteoarthritis diagnosis, which does not require radiographic evidence (age ≥ 45 years, activity-related knee pain, and no knee morning stiffness lasting >30 minutes)
* knee pain ≥ 3 months
* average pain intensity ≥ 4 on a scale from 0 to 10
* knee pain as the chief complaint
* able to understand English

Exclusion Criteria:

* current skin disease of the left ear interfering with the application of the auricular electrode for stimulation(eczema, urticarial lesion, skin infection, external otitis, etc.)
* auditory canal not adapted to the application of the ear electrode
* known history of cardiac rhythm disturbances or atrioventricular block > 1st degree, conduction disturbances
* recurrent vagal syncope
* history of vagotomy
* use of other medical devices electrically active (pacemaker, transcutaneous electrical nerve stimulation, etc)
* serious and uncontrolled concomitant disease, including cardiovascular, nervous system, pulmonary, renal, hepatic, endocrine, gastrointestinal, epileptic disease or malignant diseases
* pregnant or breastfeeding woman
* numbness or sensation loss on the body sites for pain measurements (i.e., the wrist, knee, the forearm)
* any intervention procedures for knee pain in the past 3 months
* age less than 45 years old

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-06-03 (Actual); Study Completion 2023-06-08 (Actual)

PRIMARY OUTCOMES:
Change in Pressure Pain Threshold | Same day assessment with 3 data points: baseline, immediately after- and 15 minutes after tVNS intervention
  Pressure pain thresholds (PPT) will be assessed at the wrist and patellae. PPT being assessed at a remote body site (e.g., wrist) is to measure central pain sensitivity while PPT being assessed at the location of pain (i.e., knee, patellae) is to assess peripheral pain sensitivity with or without central pain sensitivity. PPT will be assessed using a handheld pressure algometer with 1 cm2 rubber tip. PPT will be defined as the point at which the participant verbally indicated that the pressure first changed to slight pain. A lower PPT value (Kgf) represents greater pain sensitivity. PPT will be assessed 3 times at each location and averaged. Changes in PPT between immediately after tVNS and baseline and between 15 minutes after tVNS intervention and baseline will be used for analysis.
Change in Conditioned Pain Modulation | Same day assessment with 3 data points: baseline, immediately after- and 15 minutes after tVNS intervention
  Conditioned pain modulation (CPM) evaluates the adequacy of the descending pain modulatory pathways, which contributes to central pain sensitivity. Investigators will assess CPM using PPT as the test stimulus (PPT1) at the wrist as described above, with forearm ischemia using a blood pressure cuff as the conditioning stimulus. Briefly, the blood pressure cuff applied to the contralateral arm will be inflated to 10mm Hg above systolic pressure. The participant will be then instructed to perform hand grip squeezes until pain of at least 4/10 occurs in the contralateral arm. PPT will be then reassessed at the wrist 3 times and averaged (PPT2). Percent efficiency of CPM (%CPM) was computed as PPT2/PPT1, multiplied by 100; %CPM ≤ 100 indicates inefficient CPM. Changes in %CPM between immediately after tVNS intervention and baseline and between 15 minutes after tVNS intervention and baseline will be used for analysis.
Change in Temporal Summation | Same day assessment with 3 data points: baseline, immediately after- and 15 minutes after tVNS intervention
  Temporal summation (TS) is a sensitive measurement of central pain sensitivity. Investigators will assess TS using a standard set of weighted probes from 64-512 mN. Participants will rate the pain experienced by each successive weighted probe being touched on the skin of the wrist until a pain rating of ≥ 4/10 is achieved. The selected probe will be then applied at a frequency of 1 Hz for 10 seconds on the wrist. Participants will provide a pain rating at the completion of the train of 10 stimulations and 15 seconds post-stimulation. TS will be defined as the difference between the highest post-stimulation pain rating and the initial pain rating. A post-stimulation pain rating greater than the initial pain rating will be considered to be reflective of an increase in central pain sensitivity. Changes in TS between immediately after tVNS intervention and baseline and between 15 minutes after tVNS intervention and baseline will be used for analysis.
Change in Parasympathetic Function | Same day assessment with 3 data points: baseline, immediately after- and 15 minutes after tVNS intervention
  Investigators will assess changes in parasympathetic function before and immediately after- and 15 minutes after tVNS intervention. Heart rate variability (HRV), a measurement of autonomic function, will be assessed at baseline and after tVNS intervention using a wearable and wireless heart rate monitor. Investigators will have participants lie supine for 5 mins in each assessment to collect heart rate variability parameters such as high frequency and high-frequency/low-frequency ratio that is specific to activity in parasympathetic nervous system function.
Change in knee pain | Same day assessment with 3 data points: baseline, immediately after- and 15 minutes after tVNS intervention
  Investigators will assess changes in knee pain before (baseline), immediately after- and 15 minutes after tVNS intervention using a 0-10 numeric rating scale where 0 indicates no knee pain and 10 indicates the worst knee pain. Changes in knee pain between immediately after tVNS intervention and baseline and between 15 minutes after tVNS intervention and baseline will be used for analysis.
Change in and The Western Ontario McMaster Universities Osteoarthritis Index | Same day assessment with 3 data points: baseline, immediately after- and 15 minutes after tVNS intervention
  Investigators will assess changes in knee pain before (baseline), immediately after- and 15 minutes after tVNS intervention using The Western Ontario McMaster Universities Osteoarthritis Index (WOMAC). WOMAC knee pain scale ranges 0-20 with 5 questions assessing knee pain in different contexts such as knee pain during walking and pain during standing. Each question has a score of 0-4. A greater WOMAC score represents greater knee pain. Change in WOMAC score between immediately after tVNS intervention and baseline and between 15 minutes after tVNS intervention and baseline will be used for analysis.
Safety about tVNS intervention | At the end of the study visit
  Investigators will assess safety by evaluating the intervention completion rate, determined by the number of participants who completed the intervention divided by the number of participants enrolled. If there is any adverse/side effect, the types of such events will be documented.
Satisfaction Level | At the end of the study visit
  At the end of the study visit, investigators will assess the satisfaction level with tVNS intervention using the 8-item Client Satisfaction Questionnaire. The questionnaire asks about the satisfaction level regarding the new intervention using 8 questions. Each question has a 1-4 score where 1 indicates poor, and 4 indicates high satisfaction level.

SECONDARY OUTCOMES:
Pain catastrophizing scale (PCS) | Immediately before tVNS intervention
  The Pain Catastrophizing Scale is a validated 13-item scale with questions related to catastrophizing behavior. The total score is 52 with higher scores indicating greater catastrophic thoughts.
Fear avoidance belief questionnaire (FABQ) | Immediately before tVNS intervention
  The Fear-Avoidance Belief Questionnaire categorizes these traits using items related to fear about physical and work activities. A total score is 96 with 16 questions. Each item is scored from 0 to 6 with a higher number indicating increased fear of activity or work.
Pittsburgh sleep quality index (PSQI) | Immediately before tVNS intervention
  The Pittsburgh Sleep Quality Index (PSQI) is a self-reported questionnaire. PSQI contains 19 individual items, creating seven components that produce one global score, ranging from 0 to 21. A score of 0-4 indicates the absence of sleep problems, while scores 5 and higher indicate poor sleep quality.
Hospital anxiety and depression scale (HADS) | Immediately before tVNS intervention
  HADS contains seven questions about anxiety and seven questions about depression, with a 0-3 score for each question. Higher scores indicate greater anxiety and depression.
Ethnic Identity (Multigroup Ethnic Identity Measure (MEIM) | Immediately before tVNS intervention
  MEIM contains 12 questions to assess the extent to which individuals have an ethnic identity. Each question has a 1-4 score where 1 indicates poor ethnic identity and 4 indicates strong ethnic identity. Higher scores indicate that the individual has stronger feelings of belonging to the ethnic group with which he/she identified.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas at El Paso, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aoyagi K, Rivas E, Shababi R, Edwards R, LaValley M, Lechuga J, Napadow V, Neogi T. Safety and preliminary efficacy of transcutaneous auricular vagus nerve stimulation on chronic knee pain: A pilot trial. Osteoarthr Cartil Open. 2024 Nov 23;7(1):100545. doi: 10.1016/j.ocarto.2024.100545. eCollection 2025 Mar. PMID 39687279